CLINICAL TRIAL: NCT07097740
Title: A Prospective Early Feasibility Clinical Study of Surgical Implantation of a Polymer Prosthetic Heart Valve
Brief Title: Early Feasibility Study of Surgical Implantation of a Polymer Prosthetic Mitral and Aortic Valve
Acronym: POLYVALVE-FIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mitrassist Lifesciences Limited Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSVR-FIH-ZS
Record Dates: First submitted 2025-06-27; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: AORTIC VALVE DISEASES; Mitral Valve Disease; Aortic Stenosis; Aortic Regurgitation; Mitral Stenosis; Mitral Regurgitation
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Mitral Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel intervention groups:
  * Polymer Aortic Valve Replacement
  * Polymer Mitral Valve Replacement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polymer Aortic Valve Replacement (Experimental): Surgical implantation of polymer prosthetic valve in the aortic position.
  Interventions: Device: Polymer Prosthetic Heart Valve
- Polymer Mitral Valve Replacement (Experimental): Surgical implantation of polymer prosthetic valve in the mitral position.
  Interventions: Device: Polymer Prosthetic Heart Valve

INTERVENTIONS:
Device: Polymer Prosthetic Heart Valve — Surgical implantation of polymer prosthetic valve.

SUMMARY:
The goal of this clinical trial is to explore the early feasibility, initial safety, and efficacy of surgical implantation of a polymer prosthetic heart valve in patients requiring either mitral valve replacement or aortic valve replacement.

The main question it aims to answer is:

-- What is the rate of valve-related complications, including thromboembolism, valve thrombosis, severe perivalvular leak, severe bleeding, and endocarditis, at 12 months post-operation?

Participants will undergo:

* Surgical implantation of a polymer prosthetic valve (mitral valve replacement for mitral valve group and aortic valve replacement for aortic valve group).
* Regular follow-up visits at 30 days, 3-6 months, and 12 months post-operation to evaluate clinical outcomes, including echocardiographic assessment and clinical event monitoring.

DETAILED DESCRIPTION:
This is a prospective, exploratory, single-center clinical study designed to assess the early feasibility and initial safety of an investigational polymer prosthetic heart valve. A total of 10 patients will be enrolled, with 5 patients assigned to the mitral valve replacement group and 5 patients to the aortic valve replacement group.

Primary outcomes include the occurrence of valve-related complications within 12 months, such as thromboembolism, valve thrombosis, severe perivalvular leak, severe bleeding, and endocarditis.

Secondary outcomes include immediate device success rate, valve hemodynamic performance, comprehensive safety event evaluations (e.g., all-cause mortality, all-cause reoperation, valve extraction, and structural or non-structural valve dysfunction), cardiac functional classification (NYHA), and quality of life assessments (Kansas City Cardiomyopathy Questionnaire, KCCQ).

Eligible participants are patients requiring mitral or aortic valve replacement, capable of undergoing extracorporeal circulation and anticoagulation therapy, and who have provided informed consent.

Exclusion criteria include patients with prior valve replacement surgery (except transcatheter mitral valve edge-to-edge repair), urgent/emergency procedures, significant comorbidities (e.g., recent stroke or myocardial infarction, severe liver/kidney dysfunction, active infections), severe coagulation disorders, allergies to valve materials, substance abuse issues, psychiatric disorders, or anticipated life expectancy under 12 months. Patients who drop out after valve implantation will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Adults requiring surgical replacement of either mitral or aortic valve
* Capable of undergoing cardiopulmonary bypass
* Able to tolerate anticoagulation therapy
* Able to understand study purpose, willing to provide informed consent and comply with follow-up

Exclusion Criteria:

1. History of previous cardiac valve surgery or percutaneous valve replacement, including surgical aortic or mitral valve replacement (excluding Percutaneous Balloon Mitral Valvuloplasty [PBMV], which is permitted).
2. Requirement for urgent or emergency cardiac surgery.
3. Planned concurrent aortic valve surgery or combined valve procedure (e.g., simultaneous aortic and mitral valve surgery).
4. Scheduled coronary artery bypass graft (CABG) during the same admission.
5. Anticipated need for additional non-valve cardiac surgery within 12 months.
6. Active systemic infection, including pneumonia or infective endocarditis.
7. Intracardiac thrombus detected on echocardiography or imaging.
8. Stroke or transient ischemic attack within the prior 3 months.
9. Myocardial infarction, unstable coronary syndrome, or coronary revascularization within the prior 3 months.
10. Severe comorbidities with expected life expectancy <12 months, including Child-Pugh C liver disease, end-stage malignancy, or advanced pulmonary disease.
11. Participation in another interventional clinical trial involving investigational devices or drugs.
12. Anatomical risk factors such as ascending aortic aneurysm (≥50 mm), bicuspid aortic valve with ascending aorta ≥45 mm, or other high-risk features identified on imaging.
13. Left ventricular ejection fraction (LVEF) ≤35%, indicating severe systolic dysfunction.
14. Severe renal insufficiency, e.g., estimated GFR <30 mL/min/1.73 m² or requirement for chronic dialysis.
15. Coagulopathy or active bleeding disorders, e.g., INR >1.5 without anticoagulation therapy.
16. Hematologic abnormalities: hematocrit <30%, hemoglobin <100 g/L, platelet count <100 × 10⁹/L, or WBC <4 × 10⁹/L or >10 × 10⁹/L.
17. History of substance abuse, chronic alcoholism, or significant psychiatric illness impairing study compliance.
18. Preoperative or intraoperative anatomical unsuitability of the valve apparatus or cardiac structure.
19. Known allergy or hypersensitivity to polyurethane, polyester, or sulfonate-based biomaterials used in the valve prosthesis.
20. Withdrawal from the study after valve implantation (such participants are not allowed to re-enroll).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
12-Month Incidence of Valve-related Complications | 12 months post-operation
  Evaluate the incidence of valve-related complications at 12 months post-operation, including thromboembolism, valve thrombosis, severe perivalvular leak, severe bleeding, and endocarditis.

SECONDARY OUTCOMES:
Immediate Device Success Rate | Immediately post-operation
  Proportion of participants achieving successful device implantation without intraoperative complications.
Valve Hemodynamic Performance 1 Mean Transvalvular Gradient at 12 months | 12 months post-operation
  Mean pressure gradient across the valve measured by echocardiography (unit: mmHg).
Valve Hemodynamic Performance2 Effective Orifice Area (EOA) at 12 months | 12 months post-operation
  Effective orifice area of the implanted valve measured by echocardiography (unit: cm²).
Safety Outcomes and Adverse Events | Up to 12 months post-operation
  Incidence of safety-related events including all-cause mortality, all-cause reoperation, valve extraction, valve thrombosis, severe bleeding, severe perivalvular leak, structural and non-structural valve deterioration, hemolysis, endocarditis, and any other serious adverse events.
Cardiac Function Classification (NYHA) | 12 months post-operation
  Assess participants' cardiac function using New York Heart Association (NYHA) classification.
Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score at 12 months | 12 months post-operation
  Quality of life assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ).
  The KCCQ is a 23-item questionnaire measuring health status in heart failure patients, scored from 0 to 100, where higher scores indicate a better health status.
Valve Hemodynamic Performance 3 Paravalvular Leakage Severity at 12 months | 12 months post-operation
  Severity of paravalvular leakage (PVL) assessed by echocardiography, classified as None/Trace, Mild, Moderate, or Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiovascular Surgery, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided